CLINICAL TRIAL: NCT07131787
Title: Optimizing Rehabilitation After Achilles Tendon Rupture Repair: The Role of Blood Flow Restriction Training in Tendon and Muscle Recovery
Acronym: TENDON-BFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2025-0152
Record Dates: First submitted 2025-07-29; First posted 2025-08-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-04

CONDITIONS: Achilles Tendon Rupture; Blood Flow Restriction Therapy
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional therapy (Active Comparator): control group: patients in this group will undergo the same standard strength training program as the BFR-group, but without a tourniquet.
  Interventions: Other: Standardised strength training
- Blood flow restriction group (Experimental): patients in this group will undergo a standard strength training program combined with an occlusion cuff. The cuff will be used during exercises targeting quadriceps and calf muscles.
  Interventions: Device: Blood flow restriction training (smart-cuff pro device)

INTERVENTIONS:
Device: Blood flow restriction training (smart-cuff pro device) — This group will undergo low load strength training consisting of calf, thigh, glute and core exercises. A Blood flow restriction cuff will be added during selected exercises in rehabilitation program (targeting quadriceps and calf muscles)
  Other Names: Kaatsu; Partial vascular occlusion
  Arms: Blood flow restriction group
Other: Standardised strength training — This group will undergo standard, traditional strength training consisting of calf, thigh, glute and core exercises.
  Arms: Conventional therapy

SUMMARY:
The goal of this clinical trial is to investigate whether rehabilitation with blood flow restriction (BFR) offers added value compared to conventional rehabilitation in patients undergoing surgical repair for Achilles tendon rupture. The study will include adult patients of all sexes who have undergone surgical treatment at two selected hospitals.

The main questions it aims to answer are:

Does BFR-enhanced rehabilitation improve functional recovery compared to conventional rehabilitation? What are the effects of BFR on muscle strength and tendon recovery?

Researchers will compare blood flow restriction (BFR) therapy with conventional rehabilitation to determine whether BFR leads to improved clinical, muscular, and tendon-related outcomes.

Participants will:

1. Undergo standard surgical repair of the Achilles tendon
2. Be randomly assigned to a 24-week exercise therapy program-either with or without blood flow restriction (BFR)-starting four weeks post-surgery
3. Take part in follow-up assessments at weeks 4, 8, 12, 18, 24, and 52, which will include:

   * Questionnaires on pain, quality of life, fear of movement, and return to sport
   * Medical imaging techniques such as ultrasound, MRI, shear wave elastography, and power Doppler
   * Muscle strength testing
   * Blood sample collection, along with a tendon tissue sample taken during surgery

ELIGIBILITY:
Inclusion Criteria:

* patients with total midrupture Achilles tendon rupture
* surgical treatment
* > 18 years old
* able to understand and speak Dutch

Exclusion Criteria:

* Bilateral Achilles tendon rupture
* Previous Achilles tendon rupture
* Previous treatment with fluoroquinolones or cortisone
* other condition in either leg that would limit the ability to perform the exercises or evaluations
* Diabetes or rheumatic diseases
* History of deep venous thrombosis
* severe cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Achilles tendon rupture score (ATRS) | From enrollment week 0 (pre-injury score), week 12, week 18 and week 24 (the end of treatment at 6 months post-operative). Follow-up screening at week 52
  The ATRS is a validated 10-item (score 0-10) self-report questionnaire designed specifically for Achilles tendon rupture patients. total scores range from 0-100, with a higher score representing worst symptoms and physical activity.

SECONDARY OUTCOMES:
US: tendon cross-sectional area | week 4 (pre), week 8, week 12, week 18 and week 24 (post), Follow-up at week 52
  measured by ultrasound
US: tendon length | week 4 (pre), week 8, week 12, week 18 and week 24 (post), Follow-up at week 52
  Description: measured by ultrasound
SWE: tendon stiffness | week 4, week 8, week 12, week 18, week 24 Follow-up at week 52
  Tendon stiffness measured by Shear Wave Elastography, range 0-800kPa with higher kPa representing higher stiffness
Power doppler | week 4, week 8, week 12, week 18, week 24 Follow-up at week 52
  Doppler signal for vascularisation
Heel rise endurance test | week 18, week 24 Follow-up at week 52
  The Heel Rise Endurance Test (HRET) is a functional assessment used to evaluate calf muscle endurance and strength following an Achilles tendon rupture. It involves repeatedly raising up onto the toes (heel raises) on one leg until exhaustion, with the number of repetitions recorded as a measure of performance. This test helps quantify the recovery of plantar flexion strength and endurance after injury. Combined with a linear encoder, also heel rise height and work is calculated.
Possibility to perform one heel rise | week 12
  Physical test where the patient is assessed based on the ability to perform one heel rise. Yes/no
Plantarflexion strength | week 18, week 24, Follow-up at week 52
  Isokinetic strength test measured by dynamometry (Biodex)
Tampa scale of kinesophobia (TSK) | week 4, week 24
  The Tampa Scale for Kinesiophobia (TSK) is a 17-item self-report questionnaire used to assess fear of movement or re-injury (kinesiophobia) in individuals, particularly those with musculoskeletal pain. It evaluates a patient's beliefs about the potential dangers of physical activity and how those beliefs affect their willingness to move. The TSK has a 4-point Likert scale (strongly disagree to strongly agree) for each item. The total score can vary from 17 tot 68, with a higher score representing higher kinesiophobia.
EQ-5D-5L | week 0, week 4, week 12, week 24 Follow-up at week 52
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life. It consists of two parts: a descriptive system and a visual analogue scale (EQ-VAS). The descriptive system includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from "no problems" to "extreme problems" or "unable to". The EQ-VAS asks the respondent to rate their overall health on a scale of 0 to 100.
Tegner Activity Scale (TAS) | From enrollment week 0 (pre-injury), week 18, week 24, Follow-up at week 52
  The TAS is a one-item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 represents maximum disability while a level of 10 represents elite sports athletes. Patients are asked to choose the highest level of activity they partake in at that moment.
MRI: muscle volume | week 4 and week 24 (pre- and post physical therapy)
  Based on MRI images, muscle volume will be calculated of plantarflexor muscles.
MRI: fatty infiltration | week 4 and week 24 (pre- and post physical therapy)
  Based on MRI images, fatty infiltration will be calculated
Fear of rerupture | week 4, week 12, week 24 Follow-up at week 52
  Yes/no question to assess fear of rerupture of the patient
Unilateral drop jump test | week 24, Follow-up at week 52
  The drop jump test is a plyometric exercise used to assess an athlete's reactive strength, specifically their ability to quickly transition from an eccentric (lengthening) muscle contraction during landing to a concentric (shortening) contraction during jumping, also including relevance of elastic energy storage in the tendon. It involves dropping from a predetermined height and immediately jumping as high as possible upon landing. The test measures the athlete's reactive strength index (RSI), which is calculated by dividing jump height by ground contact time.
Unilateral counter movement jump | week 24, Follow-up at week 52
  A unilateral countermovement jump (CMJ) is a jump test where an individual stands on one leg and performs a countermovement before jumping as high as possible, primarily assessing single-leg explosive power and interlimb asymmetries.
International Physical Activity Questionnaire - Short form (IPAQ-SF) | week 0, week 4, week 8, week 12, week 18, week 24 Follow-up week 52
  IPAQ measures the time per week spent on walking, moderate or vigorous physical activity during different aspects of life (work, leisure, household tasks, etc.). The time active will be converted to Metabolic Equivalent of a task (MET)-minutes per week. The higher the MET value, the higher the energy expenditure/physical activity.
Tendon biopt histology | week 0
  Histologic evaluation of tendon biopt which is collected during surgery: cellularity, cell roundness (morphology), collagen arrangement and ground substance (proteogylcans).
Tendon biopt mRNA | week 0
  mRNA sequencing on tendon biopt collected during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arne Burssens, Professor, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University, Ghent, East-Flanders
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: Undecided